CLINICAL TRIAL: NCT06366620
Title: Using Peer Coaches to Extend Behavioral Parent Training Programs in Underserved Communities
Brief Title: Examining the Feasibility, Acceptability, and Fidelity of Utilizing Parent Training Graduates as Peer Supports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003416
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Child Disruptive Behavior Disorders; Parent Child Relationship; Parent Management Training; Peer Support; Child Behavior Problems; Challenging Behavior; Positive Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FAST-B PEERS (Experimental): Parents in FAST-B PEERS group will receive standard 5-week FAST-B program as well as weekly check-in support from trained 'Peer Support' parents who have previously been through parent behavioral management training programs.
  Interventions: Behavioral: FAST-B PEERS; Behavioral: FAST-B (First Approach Skills Training - Behavior)
- FAST-B (Active Comparator): Parents in FAST-B group will receive standard FAST-B program with 5 weekly group sessions with clinician.
  Interventions: Behavioral: FAST-B (First Approach Skills Training - Behavior)

INTERVENTIONS:
Behavioral: FAST-B PEERS — FAST-B PEERS consists of trained Peer Support providing weekly check-in calls with families going through FAST-B behavioral parent training program. Peer Support are parents who have previously participated in a behavioral parent training program who have undergone 6-8 hours of additional dedicated training.
  Arms: FAST-B PEERS
Behavioral: FAST-B (First Approach Skills Training - Behavior) — 5-week parent behavioral management training program

SUMMARY:
Disruptive behavioral disorders are common in early childhood, affecting up to 15% of preschool-aged children. Behavioral parent training programs are a first-line evidence-based treatment for child disruptive behaviors. There is evidence showing that (a) these programs are effective in reducing disruptive behavior and improving long-term outcomes, and (b) there is an excellent return on investment for early intervention. Nevertheless, there is limited availability of behavioral parent training programs, particularly in rural settings, due to shortages of trained clinicians. Thus, there is a pressing need for expanding the mental healthcare workforce in rural/underserved areas. The study will involve an established parent-based behavioral intervention (First Approach Skills Training for Behavior; or FAST-B) with added pilot component incorporating parents who have previously been through parent behavioral management training programs as Peer Supports.

DETAILED DESCRIPTION:
Up to 30 (15 per group, with 2 total groups) participant families will be recruited for FAST-B Peers intervention. These participants will receive the FAST-B standard of care in the context of the research study through trained clinician on the research team. As is the current standard of clinical care, FAST-B will be delivered in 1-hour weekly sessions in group-based format via Zoom, using the standard FAST-B curriculum and caregiver workbooks (https://www.seattlechildrens.org/health-safety/classes-events/behavior-basics-class/).

In addition to standard of care, half the FAST-B participants will be randomized 1:1 to additionally receive an added pilot Peer Support component. The Peer Support curriculum was developed through an iterative process, incorporating valuable feedback from parents and guidance from a dedicated community advisory panel. Upon enrollment completion of FAST-B group, randomization will be performed via random number generator. This FAST-B Peers pilot intervention involves trained Peer Supports who will each work with 2-3 families over the course of the 5-week intervention.

Peer Supports will conduct weekly calls with families going through FAST-B intervention to review the material presented, discuss application for the family, problem-solve barriers, and reinforce the family's efforts. Peer supports will additionally receive weekly consultation (1-2 hours/week) with the clinician delivering FAST-B. After the intervention is completed, both peer supports and participant families will be asked to participate in follow-up focus groups to discuss their experience in the intervention, specifically as it relates to the work of the peer supports.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child ages 3-6
* Parent has access to video-enabled device
* Parent is fluent in English or Spanish
* Child of parent has a score of at least 3 on conduct subscale of Strengths and Difficulties Questionnaire or at least 6 on hyperactivity subscale of Strengths and Difficulties Questionnaire
* Parent is comfortable being randomized to either standard intervention (FAST-B) or FAST-B with added FAST-B PEERS component.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Acceptability of FAST-B PEERS | Up to 6 weeks
  Participant rating of experience working with Peer Support, from 1 (poor) to 5 (excellent)
Acceptability of FAST-B | Up to 6 weeks
  Participant rating of FAST-B program, from 1 (poor) to 5 (excellent)
FAST-B PEERS support calls attended | Up to 6 weeks
  Percent of peer support calls attended

SECONDARY OUTCOMES:
Weekly Assessment of Child Behavior - P | Up to 6 weeks
  Standardized parent-report measure of positive child behaviors (minimum = 0; maximum = 63), with higher scores indicating higher level of positive behaviors
Coping with Child Negative Emotions Scale | Up to 6 weeks
  Standardized parent-report measure of parents typically respond to their child's negative emotions. Three subscales focus on positive responses: expressive encouragement, emotion-focused reactions, problem-focused reactions (minimum = 1 (worst), maximum = 7 (best)). Three subscales focus on negative responses: distress reactions, punitive reactions, minimization reactions (minimum = 1 (best), maximum = 7 (worst)).
Strengths and Difficulties Questionnaire | Up to 6 weeks
  Standardized measurement of child strengths and difficulties across behavioral domains, yielding Total Difficulties Score (minimum = 0 (best); maximum = 40 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Julia T Mattson, MD, PhD, Principal Investigator — Seattle Children's/University of Washington; Alissa D Hemke, MD, Principal Investigator — Seattle Children's/University of Washington
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Recordings of behavioral intervention sessions, peer support calls, and post-intervention focus groups will not be shared with anybody outside of approved research team members involved in coding process. Data from the pilot intervention will be shared in conference abstracts and peer-reviewed journal publications.